CLINICAL TRIAL: NCT06501755
Title: Effects and Mechanisms of Action of an Individualized Theta Frequency Transcranial Alternating Current Stimulation (ITF-tACS) on a Working Memory Training at Healthy Older Adults With Subjective Cognitive Decline (SCD)
Brief Title: Effects of Individualized Theta-tACS on a Working Memory Training at SCD
Acronym: tACOSenior
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: tACOSenior
Record Dates: First submitted 2024-06-27; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-04

CONDITIONS: Subjective Cognitive Decline
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham tACS (Sham Comparator): Intensity: 2 mA (peak-to-peak), localisation: F4/P4, phase-shift between the electrodes: 0°,duration: 20s at the begin and the end of the task (adaptive spatial n-back) with additionally each time 15 s fade-in and fade-out, frequency: 6Hz.
  Interventions: Device: transcranial alternating current stimulation (tACS)
- Individualized Theta-Frequency tACS (Experimental): Intensity: 2 mA (peak-to-peak), localisation: F4/P4, phase-shift between the electrodes: 0°, duration: 27 min with 15 s fade-in and fade-out, frequency: peak theta-frequency at the baseline measurement during the execution of the spatial 2-, 3-, and 4-back.
  Interventions: Device: transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: transcranial alternating current stimulation (tACS) — Transcrainal alternating current stimulation (tACS) is a non-invasive brain-stimulation where weak sinusoidal electric current with frequencies within the EEG-range is applied over electrodes on the scalp. In the study we use the DC-Stimulator MC, neuroConn, Ilmenau for the stimulation.The device is authorized as medical device for the application on humans in Germany with a CE-Identification. We use two circular (area each = ca. 7.07 cm^2) and two ring-shaped (area each = 40 cm^2) rubber electrodes. Impedances are kept < 15 kOhm.

SUMMARY:
The aim of the study is to investigate the effects and mechanisms of action of an individualized transcranial alternating current stimulation in the theta-range (ITF-tACS) on a three day spatial working memory training in healthy older adults with subjective cognitive decline (SCD).

DETAILED DESCRIPTION:
This study uses a randomized, double-blind, two-armed, sham-controlled between-subjects design. It is conducted at the University Hospital for Psychiatry and Psychotherapy Tübingen, Germany. Participants older than 60 years and with subjective cognitive decline (SCD) will be included. Other inclusion and exclusion criteria are displayed under "Eligibility". Participants are recruited via email-newsletters at the University of Tübingen, flyers and newspaper advertisement. Participants will receive financial compensation. A stratified block randomization is applied after the inclusion of the participants and before the baseline-session. The person generating the randomization list is not involved with data collection. Operators do not have access to the randomization list during the data collection.

Sample size is N = 36 with n = 18 participants in each group. As a phase 2 study, the aim of this study is the determination of effect sizes which can be used for further investigations. Thus due to a lack of comparable studies, no power analysis could be conducted. The group size is therefore based on the most frequently found group size (n = 18) observed in a systematic review regarding the effects of tACS targeting the memory in healthy adults.

The study includes seven time points: screening-session, baseline-session (in the end of the first week of data-collection), three training sessions (within the second week of data-collection, each session two days apart), post-session (10-12 days after the baseline-session; in the beginning of the third week of data-collection) and follow-up session (one month after the post-session). Online tACS is applied during the training sessions while the participants will conduct an adaptive spatial n-back task (online stimulation). Resting-state EEG as well as EEGs during the spatial 2-, 3-, 4-back at the baseline- and the post-session are conducted. Two groups are compared: one group with individualized theta-tACS (ITF-tACS) and one with sham-tACS.

Hypothesis H1 contains the effect on the trained task (spatial 2-, 3-, 4-back) at the post-session. The investigators expect a higher performance in the group with ITF-tACS compared to sham-tACS. To test this hypothesis, two ANCOVAs (dependent variable = performance at post-session (Reaction time and d prime, Covariate = performance at baseline-session) will be conducted.

Hypothesis H2.1 contains the effect on the trained task in the training sessions concurrent to the tACS. The investigators expect a higher performance in the group with ITF-tACS compared to sham-tACS in all sessions. To test the hypothesis, a linear mixed model will be conducted.

Hypothesis H2.2 contains the long-term effect on the trained task at the follow-up session. The investigators expect a higher performance in the group with ITF-tACS compared to sham-tACS. To test the hypothesis, two ANCOVAs will be conducted.

Hypothesis H2.3 contains the transfer effects on the verbal working memory (digit span task) at the post-session. The investigators expect a higher performance in the group with ITF-tACS compared to sham-tACS. To test the hypothesis, three ANCOVAs will be conducted.

Hypothesis H2.4 contains the effect of the training on the subjective cognitive decline (10-point Likert-scale) at the post-session. The investigators expect a lower scoring in the group with ITF-tACS compared to sham-tACS. To test the hypothesis, an ANCOVA will be conducted.

Hypothesis H2.5 contains the effect of neurophysiological measures of the spatial working memory (EEG). The investigators expect a higher theta-power and fronto-parietal connectivity in the group with ITF-tACS compared to sham-tACS.

Exploratively measures for the accuracy in the trained task, transfer effect at follow-up session for the transfer task, subjective cognitive decline (subjective cognitive decline questionnaire), quality of live (WHO-5), side effects and for sleep (Karolinska sleepiness scale, Insomnia Severity Index) are evaluated.

For all analyses the alpha level for significance is set to p < 0.05. Because reaction times < 150 ms are regarded as unintended and > mean reaction time + 3 SD per participant are regarded as additionally including different processes than only working memory, reaction times < 150 ms and > mean reaction time + 3 SD per participant per session are excluded from the analyses. Participants who did not complete the post-session or will miss > 1/3 of the training sessions are excluded from analyses. We test model assumptions in all analyses and control for multiple testing in the primary analyses. An interim analysis is conducted in 09/2024.

The study will provide important implications for the usage of multi-session ITF-tACS in the context of healthy aging.

ELIGIBILITY:
Inclusion Criteria:

* age >/= 60 years
* subjective cognitive decline with a duration > 6 month and without a concrete cause
* right-handedness (score > 48 in the Edinburgh Handedness Inventory (EHI; Oldfield, 1971))
* corrected or sufficient eyesight
* sufficient knowledge in German
* ability to consent

Exclusion Criteria:

* neuropsychiatric diagnose
* score > 13 in the DemTect (Kalbe et al., 2019)
* score > 4 in the Geriatric Depression Scale Short Form (GDS-SF; Sheikh & Yesavage, 1986)
* score > 16 Geriatric Anxiety Scale German version(GAS-G; Gottschling et al., 2016)
* substance abuse or dependence
* epileptic seizure in medical history
* metall in skalp-area
* pacemaker
* gravidity
* psychiatric medication
* benzodiazepines in a dosage > 1 mg Lorazepam
* participation in a tACS in history

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-07-19 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Reaction time in the spatial 2-, 3-, 4-back at the post-session | Post-session (10-12 days after the baseline-session)
  Reaction times < 150ms and > M + 3 SD after visual inspection via histogram and box plot per participant will be excluded from the analysis
d prime in the spatial 2-, 3-, 4-back at the post-session | Post-session (10-12 days after the baseline-session)
  d prime = z(Hits) - z(False Alarms)

SECONDARY OUTCOMES:
Reaction time in the adaptive spatial n-back during the trainingssessions | Trainingssessions (conducted in the week after the baseline-session with each 2 days apart)
  Reaction times < 150ms and > M + 3 SD after visual inspection via histogram and box plot per participant will be excluded from the analysisfrom the analysis
Reaction time in the spatial 2-, 3-, 4-back at the follow-up session | Follow-up session (1 month after the post-session)
  Reaction times < 150ms and > M + 3 SD after visual inspection via histogram and box plot per participant will be excluded from the analysis
d prime in the spatial 2-, 3-, 4-back at the follow-up session | Follow-up session (1 month after the post-session)
  d prime = z(Hits) - z(False Alarms)
Score on a 10-point likert scale about the worries on cognitive abilities at the post-session | Post-session (10-12 days after the baseline-session)
  The task of the participant is to rate the extend of worries about their cognitive abilities on a ten-stage scale from "no worries" to "very strong worries". With higher scores indicating stronger worries.
Sumscores in the digit span task at the post-session | Post-session (10-12 days after the baseline-session)
Theta-power in the EEG at the post-session | Post-session (10-12 days after the baseline-session)
Connectivity of the front-parietal network in the EEG at the post-session | Post-session (10-12 days after the baseline-session)

OTHER OUTCOMES:
Sumscores in the digit span task at the follow-up session | Follow-up session (1 month after the post-session)
Score on a 10-point likert scale about the worries on cognitive abilities at the follow-up session | Follow-up session
  The task of the participant is to rate the extend of worries about their cognitive abilities on a ten-stage scale from "no worries" to "very strong worries". With higher scores indicating stronger worries.
Score in the WHO-5 (Topp et al., 2015) in the post-session | Post-session (10-12 days after the baseline-session)
  The task of the participants is to rate 5 items on a six-stage scale from "all of the time" to "at non time". With higher scores indicating a higher quality of life.
Score in the WHO-5 (Topp et al., 2015) in the follow-up session | Follow-up session (1 month after the post-session)
  The task of the participants is to rate 5 items on a six-stage scale from "all of the time" to "at non time". With higher scores indicating a higher quality of life.
Score in the Insomnia Severity Index (Morin, 1993) in the post-session | post-session (10-12 days after the baseline-session)
  The task of the participants is to rate 7 items on a five-stage scale from "not at all" to "very strong" for items 1 to 3, on a scale from "very satisfied" to "very dissatisfied" for item 4 and on a scale from "not at all" to "very strong" for items 5 to 7. With higher scores indicating a stronger impairment in the sleep.
Score in the Insomnia Severity Index (Morin, 1993) in the follow-up session | Follow-up session (1 month after the post-session)
  The task of the participants is to rate 7 items on a five-stage scale from "not at all" to "very strong" for items 1 to 3, on a scale from "very satisfied" to "very dissatisfied" for item 4 and on a scale from "not at all" to "very strong" for items 5 to 7. With higher scores indicating a stronger impairment in the sleep.
Score in the Subjective Cognitive Decline Questionnaire (Rami et al., 2014) in the post-session | Post-session (10-12 days after the baseline-session)
  The task of the participants is to either to agree ("yes") or disagree ("no") to 24 items regarding their self-perceived cognitive decline over the last two years (MyCog). With higher scores indicating a stronger self-perceived cognitive decline.
Score in the Subjective Cognitive Decline Questionnaire (Rami et al., 2014) in the follow-up session | Follow-up session (1 month after the post-session)
  The task of the participants is to either to agree ("yes") or disagree ("no") to 24 items regarding their self-perceived cognitive decline over the last two years (MyCog). With higher scores indicating a stronger self-perceived cognitive decline.
Score in the Karolinska Sleepiness Scale (Akerstadt & Gillberg, 1990) after the trainingssessions | Trainingssessions (conducted in the week after the baseline-session with each 2 days apart)
  The task of the participants is to rate 5 items on a ninge-stage scale from "extremely awake" to "Very sleepy, can only stay awake with great difficulty; fight against sleep". With higher scores indicating a higher degree of sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Christian Plewnia, Principal Investigator — Universitätsklinik für Psychiatrie und Psychotherapie Tübingen, Tübingen, DE
Locations (1):
- Universitätsklinik für Psychiatrie und Psychotherapie Tübingen, Neurophysiologie & Interventionelle Neuropsychiatrie, Tübingen, DE, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Akerstedt T, Gillberg M. Subjective and objective sleepiness in the active individual. Int J Neurosci. 1990 May;52(1-2):29-37. doi: 10.3109/00207459008994241. PMID 2265922
- [Background] Gottschling, J, Segal, D. L., Häusele C., Spinath, F. M., & Stoll, G. Assessment of Anxiety in Older Adults: Translation and Psychometric Evaluation of the German Version of the Geriatric Anxiety Scale (GAS). Journal of Psychopathology and Behavior Assessment. 2016; 38: 136-148. doi: 10.1007/s10862-015-9504-z
- [Background] Kalbe, E., Calabrese, P., & Kessler, J. (2019). DemTect® Zur Unterstützung der Demenz-Diagnostik (1. Auflage.). Hogrefe.
- [Background] Morin, C.M. (1993). Insomnia: Psychological assessment and management. Guilford Press.
- [Background] Rami L, Mollica MA, Garcia-Sanchez C, Saldana J, Sanchez B, Sala I, Valls-Pedret C, Castellvi M, Olives J, Molinuevo JL. The Subjective Cognitive Decline Questionnaire (SCD-Q): a validation study. J Alzheimers Dis. 2014;41(2):453-66. doi: 10.3233/JAD-132027. PMID 24625794
- [Background] Sheikh, R.L. & Yesavage, J.A. Geriatric Depression Scale (GDS). Clinical Gerontologist. 1986; 5: 165-173.
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Booth SJ, Taylor JR, Brown LJE, Pobric G. The effects of transcranial alternating current stimulation on memory performance in healthy adults: A systematic review. Cortex. 2022 Feb;147:112-139. doi: 10.1016/j.cortex.2021.12.001. Epub 2021 Dec 24. PMID 35032750